CLINICAL TRIAL: NCT00889772
Title: Identifying Patients at Risk of Acute Lung Injury (ALI) and Acute Respiratory Distress Syndrome (ARDS) at the Time of Hospital Admission: External Validation of a Lung Injury Prediction Score (LIPS)
Brief Title: Lung Injury Prediction Study
Acronym: USCTG-LIPS1
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Temple University (Other); Johns Hopkins University (Other); University of Medicine and Dentistry of New Jersey (Other); University of Colorado, Denver (Other); University of Pennsylvania (Other); Brigham and Women's Hospital (Other); Boston University (Other); University of Michigan (Other); University of Texas Southwestern Medical Center (Other); Providence Health & Services (Other); University of Illinois at Chicago (Other); Wake Forest University (Other); Bridgeport Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Wright State University (Other); University of Missouri-Columbia (Other); Uludag University (Other); Akdeniz University (Other)
Responsible Party: Principal Investigator, Ognjen Gajic, Consultant - Critical Care, Mayo Clinic
Other Study IDs: 08-008726; USCIITG-LIPS1
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2012-06

CONDITIONS: Respiratory Distress; Acute Lung Injury
Keywords: Respiratory distress, adult; risk; emergency room; high risk surgery; sepsis; trauma; aspiration; pneumonia
MeSH Terms: conditions — Dyspnea; Acute Lung Injury; Emergencies; Sepsis; Wounds and Injuries; Pneumonia

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to externally validate the acute lung injury/acute respiratory distress syndrome (ALI/ARDS) prediction model (Lung Injury Prediction Score - LIPS) in a multicenter sample of patients at risk presented to the acute care hospitals: United States Critical Illness and Injury Trials Group (USCIITG).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult patients with one of the known risk factors for acute lung injury at the time of hospital admission

Exclusion Criteria:

* ALI/ARDS already present at the time of hospital admission, denied use of medical records for research, children, hospital readmission, transfer from another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients >18 years of age with one or more predisposing conditions for ALI/ARDS (pneumonia, sepsis, shock, pancreatitis, aspiration, high risk trauma and high risk surgery) at the time of hospital admission
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Acute Lung Injury or Acute Respiratory Distress Syndrome | during hospital stay

SECONDARY OUTCOMES:
Survival | in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Ognjen Gajic, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] George N, Elie-Turenne MC, Seethala RR, Baslanti TO, Bozorgmehri S, Mark K, Meurer D, Bihorac A, Aisiku IP, Hou PC; U.S. Critical Illness and Injury Trials Group-Lung Injury Prevention Study Investigators. External Validation of the qSOFA Score in Emergency Department Patients With Pneumonia. J Emerg Med. 2019 Dec;57(6):755-764. doi: 10.1016/j.jemermed.2019.08.043. Epub 2019 Nov 15. PMID 31735660
- [Derived] Chang SY, Dabbagh O, Gajic O, Patrawalla A, Elie MC, Talmor DS, Malhotra A, Adesanya A, Anderson HL 3rd, Blum JM, Park PK, Gong MN; United States Critical Illness and Injury Trials Group: Lung Injury Prevention Study Investigators (USCIITG-LIPS). Contemporary ventilator management in patients with and at risk of ALI/ARDS. Respir Care. 2013 Apr;58(4):578-88. doi: 10.4187/respcare.01755. PMID 22906363
- [Derived] Gajic O, Dabbagh O, Park PK, Adesanya A, Chang SY, Hou P, Anderson H 3rd, Hoth JJ, Mikkelsen ME, Gentile NT, Gong MN, Talmor D, Bajwa E, Watkins TR, Festic E, Yilmaz M, Iscimen R, Kaufman DA, Esper AM, Sadikot R, Douglas I, Sevransky J, Malinchoc M; U.S. Critical Illness and Injury Trials Group: Lung Injury Prevention Study Investigators (USCIITG-LIPS). Early identification of patients at risk of acute lung injury: evaluation of lung injury prediction score in a multicenter cohort study. Am J Respir Crit Care Med. 2011 Feb 15;183(4):462-70. doi: 10.1164/rccm.201004-0549OC. Epub 2010 Aug 27. PMID 20802164
- [Derived] Trillo-Alvarez C, Cartin-Ceba R, Kor DJ, Kojicic M, Kashyap R, Thakur S, Thakur L, Herasevich V, Malinchoc M, Gajic O. Acute lung injury prediction score: derivation and validation in a population-based sample. Eur Respir J. 2011 Mar;37(3):604-9. doi: 10.1183/09031936.00036810. Epub 2010 Jun 18. PMID 20562130